CLINICAL TRIAL: NCT07311837
Title: Investigating the Relationships Between Body Composition, Waist/Hip Ratio, Peripheral Muscle Strength, and Cough Force in Healthy Young Adults
Brief Title: Investigating the Relationships Between Body Composition, Peripheral Muscle Strength, and Cough Force in Healthy Young Adults
Status: Not yet recruiting | Type: Observational
Sponsor: Nigde Omer Halisdemir University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, Nazire Nur YILDIZ, P.T., Ph.D., Nigde Omer Halisdemir University
Other Study IDs: 2025/09-10-TUBITAK 2209-A
Record Dates: First submitted 2025-11-18; First posted 2025-12-31 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Healthy Young Adults
Keywords: Body composition; Waist-to-hip ratio; Peripheral muscle strength; Peak expiratory flow; Cough strength

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy Young Adults: Healthy individuals between the ages of 18 and 30 who volunteer to participate in the study will be included in the study.

SUMMARY:
Introduction: Body mass index (BMI) is a key parameter used for obesity classification and the evaluation and monitoring of individuals' health status. Obesity, described by the World Health Organization as a major global epidemic, remains one of the most significant preventable and manageable conditions contributing to increased risks of cardiovascular and metabolic diseases. In addition to BMI, anthropometric measurements such as the waist-to-hip ratio are crucial indicators for risk assessment. While numerous studies in the literature have addressed the detrimental effects of obesity on respiratory functions, no study has specifically examined the relationship between cough strength-a vital respiratory parameter that reflects expiratory muscle strength- and body composition, waist-to-hip ratio, and peripheral muscle strength. Furthermore, although several studies have investigated the association between grip strength-a recognized indicator of peripheral muscle function in healthy individuals-and cough strength, no research to date has explored the relationship between pinch grip strength and cough strength.

Objective: This study aims to investigate the relationships among body composition, waist-to-hip ratio, peripheral muscle strength, and cough strength in healthy young adults.

Methods: This study was designed as a cross-sectional analysis. After providing detailed information about the study to potential participants, written informed consent will be obtained in duplicate from those who agree to participate. Following the completion of a general assessment form that captures demographic characteristics, each participant's height will be measured using a measuring tape. Body composition parameters-including body weight, BMI, body fat percentage, total body water percentage, muscle mass, basal metabolic rate, and metabolic age-will be assessed using a bioelectrical impedance analysis device (Tanita) available at our faculty.

Waist and hip circumferences will be measured and used to calculate the waist-to-hip ratio for each participant. Peripheral muscle strength will be assessed using a hydraulic hand dynamometer and a pinch meter, while cough strength will be evaluated using a peak cough expiratory flow meter (PEF meter). All measurements will be repeated three times, with the best result recorded for analysis. Results: Statistical analysis will be performed using IBM SPSS Statistics version 30 (SPSS Inc., Chicago, IL, USA). Normality of continuous variables will be assessed through normality tests, coefficient of variation, and graphical representations (e.g., histograms, detrended plots). Descriptive statistics will be presented as mean ± standard deviation for normally distributed variables, and as median and interquartile range for non-normally distributed variables. Categorical variables will be expressed as percentages (%). Pearson correlation analysis will be used for normally distributed variables, and Spearman correlation analysis for non-normally distributed ones. The appropriate correlation coefficients and p-values will be reported. A p-value of <0.05 will be considered statistically significant.

Discussion: Interpretation will be based on the results of the statistical analyses.

DETAILED DESCRIPTION:
Body mass index (BMI) is an important parameter used to assess and monitor the health status of individuals by classifying obesity. Obesity, defined as a major epidemic by the World Health Organization, is the most important preventable and controllable problem that increases the risk of cardiovascular and metabolic diseases. It is estimated that more than 1 billion adults worldwide will be obese by 2030 (1,2). The COVID-19 pandemic and the increasing dependence on technology are increasing the sedentary population and changing dietary habits, thereby increasing obesity rates (3,4). In addition to BMI, the waist-to-hip ratio, an anthropometric measurement, is also an important parameter in determining risk. In individuals with abdominal fat or atrophy in large muscle groups, waist circumference may be larger than hip circumference. This results in a high waist-to-hip ratio (5). Many studies conducted during the COVID-19 pandemic have reported higher COVID-19-related mortality rates in countries with obese or overweight individuals. This situation has revealed that overweight and obese individuals are a highly vulnerable group to epidemic diseases (1). Furthermore, the literature has addressed the mechanical effects of obesity on the respiratory system, and its relationship with asthma and other respiratory diseases has been discussed (6,7). It has been reported that all respiratory function parameters are negatively affected in obese individuals with a high BMI, and other physiological mechanisms affecting respiratory mechanics are not yet understood (8-11). It is known that the abdominal muscles, which are active during forced expiration, are associated with cough force, a forced expiratory maneuver. It is thought that cough force will decrease with increasing BMI and obesity, along with weakening of the abdominal wall muscles and abdominal fat accumulation. While there are studies in the literature mentioning the negative effects of obesity on respiratory function and reporting that grip strength is related to cough force in healthy individuals (12), no studies have been found on the relationship between cough force, an important respiratory parameter that reflects expiratory muscle strength, and body composition, waist/hip ratio, and peripheral muscle strength. Our study will be the first and pioneering study to investigate the relationships between body composition, waist-to-hip ratio, peripheral muscle strength, and cough strength in healthy young adults. Furthermore, the fact that body composition will be measured using the body analysis system, the gold standard method, increases the originality of our study. One of the unique merits of our study is that it will reveal the relationships between body composition, waist-to-hip ratio, peripheral muscle strength, and cough strength in individuals known to be healthy and free of chronic diseases.

ELIGIBILITY:
Inclusion Criteria:

* Individuals between the ages of 18-30 who volunteered to participate in the study

Exclusion Criteria:

* Individuals who have a serious orthopedic, neurological or systemic disease that would prevent participation in the study and who do not volunteer to participate in the study

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy young individuals
Sampling Method: Probability Sample
Enrollment: 46 (Estimated)
Dates: Start 2026-02-15 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-15 (Estimated)

PRIMARY OUTCOMES:
Body weight | Baseline
  It expresses body weight in kilograms.
Body mass index | Baseline
  Body weight (kg) divided by the square of height (m2)
Body fat ratio | Baseline
  A measure of body fat in percent (%).
Body fluid ratio | Baseline
  A measure of the amount of fluid in the body expressed as a percentage (%).
Muscle ratio | Baseline
  The measure that expresses the lean body weight, that is, the muscle ratio in the body.
Basal metabolic rate | Baseline
  It is defined as the amount of calories the body burns while performing its basic, basal life-sustaining function (kcal and kj)
Metabolic age | Baseline
  Metabolic age is a measure of how efficiently your body's metabolism works compared to other individuals in your age group (years).
Cough strength | Baseline
  Cough strength is the measure that expresses peak-expiratory flow (PEF) during cough. It is measured with a PEF-meter.

SECONDARY OUTCOMES:
Waist-hip ratio | Baseline
  It is the result measure expressing the ratio of waist circumference measurement (cm) to hip circumference measurement (cm).
Handgrip strength | Baseline
  Handgrip strength (HGS) is a simple and reliable measurement of maximum voluntary muscle strength. It is defined as an index of upper limb strength and functional recovery, measured using tools like the dynamometer, which is considered the gold standard for its reliability and validity.
Pinch strength | Baseline
  Pinch strength refers to the force exerted during precision grasp activities, specifically when the thumb tip contacts the tip of one or more fingers, such as in two-point pinch or three-point pinch configurations. It is a critical component of hand function that involves the coordinated action of the thumb and fingers.

CONTACTS AND LOCATIONS:
Overall Officials: Nazire Nur YILDIZ, Ph.D., Study Chair — Nigde Omer Halisdemir University
Locations (1):
- Nigde Omer Halisdemir University, Faculty of Bor Health Sciences, Niğde, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Since the work has not started yet, it cannot be shared.

REFERENCES:
- [Background] Mafort TT, Rufino R, Costa CH, Lopes AJ. Obesity: systemic and pulmonary complications, biochemical abnormalities, and impairment of lung function. Multidiscip Respir Med. 2016 Jul 12;11:28. doi: 10.1186/s40248-016-0066-z. eCollection 2016. PMID 27408717